CLINICAL TRIAL: NCT05583396
Title: Pulmonary Diffusing Capacity to Nitric Oxide and Carbon Monoxide During Exercise in Patients With Chronic Obstructive Pulmonary Disease: a Test-retest Reliability Study
Brief Title: Pulmonary Diffusing Capacity During Acute Exercise in Patients With COPD
Acronym: DiffLung2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Ronan Berg, MD, DMSc, Associate Professor, Principal investigator, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DiffLung2
Record Dates: First submitted 2022-10-13; First posted 2022-10-17 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Pulmonary diffusing capacity; Reliability; Test-retest
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acute exercise (Other): Pulmonary diffusing capacity using the DLCO/NO technique is assessed at rest and during exercise (60% of maximal workload on a bicycle ergometer)
  Interventions: Diagnostic Test: Acute exercise

INTERVENTIONS:
Diagnostic Test: Acute exercise — The measurement will be repeated within one to seven days.

SUMMARY:
The combined measurement of the pulmonary diffusing capacity to carbon monoxide (CO) and nitric oxide (NO) (DLCO/NO) during exercise may be a useful physiological measure of alveolar-capillary reserve in patients with Chronic obstructive pulmonary disease (COPD). The present study investigated the test-retest reliability of DLCO/NO-based metrics.

DETAILED DESCRIPTION:
The combined measurement of the pulmonary diffusing capacity to carbon monoxide (CO) and nitric oxide (NO) (DLCO/NO) has recently been standardised and validated for clinical use. It is thus ideal for assessing acute changes in pulmonary diffusing capacity and its components during various physiological manoeuvres. These changes are thought to involve acute changes in pulmonary perfusion and are notably relevant for patients with chronic obstructive pulmonary disease (COPD), in which they may be related to exertional dyspnoea. The aim of the present study is to investigate the effects of acute exercise on pulmonary diffusing capacity, and to determine the day-to-day repeatability of such assessments.

ELIGIBILITY:
Inclusion Criteria:

* Chronic obstructive pulmonary disease (GOLD II + III)

Exclusion Criteria:

* Known heart disease
* Pregnancy
* Disease within two weeks prior to inclusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Rest-to-exercise change in DLNO | Measured at day 1 and day 2
  The physiological change from rest to exercise in DLNO obtained using the combined DLCO/NO technique with a 5-sec breathhold.
Rest-to-exercise change in DLCOc | Measured at day 1 and day 2
  The physiological change from rest to exercise in DLCOc obtained using the combined DLCO/NO technique with a 5-sec breathhold.
Rest-to-exercise change in DM | Measured at day 1 and day 2
  The physiological change from rest to exercise in DM obtained using the combined DLCO/NO technique with a 5-sec breathhold.
Rest-to-exercise change in VC | Measured at day 1 and day 2
  The physiological change from rest to exercise in VC obtained using the combined DLCO/NO technique with a 5-sec breathhold.
Rest-to-exercise change in VA | Measured at day 1 and day 2
  The physiological change from rest to exercise in VA obtained using the combined DLCO/NO technique with a 5-sec breathhold.
Smallest real difference (SRD) for Diffusion capacity for DLNO at rest | Measured at day 1 and day 2
  SRD with 95 % confidence intervals (95% CI) for DLNO at rest
SRD for DLNO during exercise | Measured at day 1 and day 2
  SRD with 95% CI for DLNO during exercise
SRD for Diffusion capacity for carbon monoxide (DLCOc) at rest | Measured at day 1 and day 2
  SRD with 95% CI for DLCOc at rest
SRD for DLCOc during exercise | Measured at day 1 and day 2
  SRD with 95% CI for DLCOc during exercise
SRD for membrane diffusing capacity (DM) at rest | Measured at day 1 and day 2
  SRD with 95% CI for DM at rest
SRD for DM during exercise | Measured at day 1 and day 2
  SRD with 95% CI for DM during exercise
SRD for Pulmonary blood volume (Vc) at rest | Measured at day 1 and day 2
  SRD with 95% CI for Vc at rest
SRD for Vc during exercise | Measured at day 1 and day 2
  SRD with 95% CI for Vc during exercise
SRD for alveolar volume (VA) at rest | Measured at day 1 and day 2
  SRD with 95 % CI for VA at rest
SRD for VA during exercise | Measured at day 1 and day 2
  SRD with 95 % CI for VA during exercise
Coefficient of Variance (CV) for DLNO at rest | Measured at day 1 and day 2
  CV with a 95% CI at rest
CV for DLNO during exercise | Measured at day 1 and day 2
  CV with a 95% CI during exercise
CV for DLCOc at rest | Measured at day 1 and day 2
  CV with 95% CI for DLCOc at rest
CV for DLCOc during exercise | Measured at day 1 and day 2
  CV with 95% CI for DLCOc during exercise
CV for DM at rest | Measured at day 1 and day 2
  CV with 95% CI for DM at rest
CV for DM during exercise | Measured at day 1 and day 2
  CV with 95% CI for DM during exercise
CV for Vc at rest | Measured at day 1 and day 2
  CV with 95% CI for DM at rest
CV for Vc during exercise | Measured at day 1 and day 2
  CV with 95% CI for DM during exercise
CV for VA at rest | Measured at day 1 and day 2
  CV with 95% CI for VA at rest
CV for VA during exercise | Measured at day 1 and day 2
  CV with 95% CI for VA during exercise
Intraclass correlation coefficient (ICC) for DLNO at rest | Measured at day 1 and day 2
  ICC for DLNO with 95% CI at rest
Intraclass correlation coefficient (ICC) for DLNO during exercise | Measured at day 1 and day 2
  ICC for DLNO with 95% CI during exercise
ICC for DLCOc at rest | Measured at day 1 and day 2
  ICC for DLCOc with 95% CI at rest
ICC for DLCOc during exercise | Measured at day 1 and day 2
  ICC for DLCOc with 95% CI during exercise
ICC for DM at rest | Measured at day 1 and day 2
  ICC for DM with 95% CI at rest
ICC for DM during exercise | Measured at day 1 and day 2
  ICC for DM with 95% CI during exercise
ICC for VC at rest | Measured at day 1 and day 2
  ICC for VC with 95% CI at rest
ICC for VC during exercise | Measured at day 1 and day 2
  ICC for VC with 95% CI during exercise
ICC for VA at rest | Measured at day 1 and day 2
  ICC for VA with 95% CI at rest
ICC for VA during exercise | Measured at day 1 and day 2
  ICC for VA with 95% CI during exercise

SECONDARY OUTCOMES:
Diffusion capacity for nitric oxide (DLNO) at rest | Measured at day 1 and day 2
  DLNO at rest obtained using the combined DLCO/NO technique with a 5-sec breathhold.
Diffusion capacity for nitric oxide (DLNO) during exercise | Measured at day 1 and day 2
  DLNO during exercise obtained using the combined DLCO/NO technique with a 5-sec breathhold.
Diffusion capacity for carbon monoxide (DLCOc) at rest | Measured at day 1 and day 2
  DLCOc at rest obtained using the combined DLCO/NO technique with a 5-sec breathhold.
Diffusion capacity for carbon monoxide (DLCOc) during exercise | Measured at day 1 and day 2
  DLCOc during exercise obtained using the combined DLCO/NO technique with a 5-sec breathhold.
Membrane diffusing capacity (DM) at rest | Measured at day 1 and day 2
  DM at rest obtained using the combined DLCO/NO technique with a 5-sec breathhold.
Membrane diffusing capacity (DM) during exercise | Measured at day 1 and day 2
  DM during exercise obtained using the combined DLCO/NO technique with a 5-sec breathhold.
Pulmonary blood volume (Vc) at rest | Measured at day 1 and day 2
  VC at rest obtained using the combined DLCO/NO technique with a 5-sec breathhold.
Pulmonary blood volume (Vc) during exercise | Measured at day 1 and day 2
  VC during exercise obtained using the combined DLCO/NO technique with a 5-sec breathhold.
Breath hold time at rest | Measured at day 1 and day 2
  Breath hold time at rest obtained using the combined DLCO/NO technique with a 5-sec breathhold.
Breath hold time during exercise | Measured at day 1 and day 2
  Breath hold time during exercise obtained using the combined DLCO/NO technique with a 5-sec breathhold.
Alveolar volume (VA) at rest | Measured at day 1 and day 2
  VA at rest obtained using the combined DLCO/NO technique with a 5-sec breathhold.
Alveolar volume (VA) during exercise | Measured at day 1 and day 2
  VA during exercise obtained using the combined DLCO/NO technique with a 5-sec breathhold.
Bland Altman Plot - DLNO | Measured at day 1 and day 2
  Bland Altman plot for repeated measures for DLNO
Bland Altman Plot - DLCOc | Measured at day 1 and day 2
  Bland Altman plot for repeated measures for DLCOc
Bland Altman Plot - DM | Measured at day 1 and day 2
  Bland Altman plot for repeated measures for DM
Bland Altman Plot - VC | Measured at day 1 and day 2
  Bland Altman plot for repeated measures for VC
Bland Altman Plot - VA | Measured at day 1 and day 2
  Bland Altman plot for repeated measures for VA

OTHER OUTCOMES:
Forced Expiratory Volume in 1 second (FEV1) | Measured at baseline
  FEV1 measured during dynamic spirometry, and expressed as liter and percentage of predicted.
Forced vital capacity (FVC) | Measured at baseline
  FVC measured during dynamic spirometry, and expressed as liter and percentage of predicted.
FEV1/FVC ratio | Measured at baseline
  FEV1/FVC measured during dynamic spirometry, and expressed as liter and percentage of predicted.
Residual Volume (RV) | Measured at baseline
  RV measured with whole-body plethysmography, and expressed as liter and percentage of predicted.
Total Lung Capacity (TLC) | Measured at baseline
  TLC measured with whole-body plethysmography, and expressed as liter and percentage of predicted.
Diffusion capacity for carbon monoxide corrected for hemoglobin | Measured at baseline
  DLCOc measured and expressed as mmol/(min*kPa) and percentage of predicted.
Peak oxygen consumption (VO2peak) | Measured at baseline
  VO2peak test performed on a Monark ergometer bicycle.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Centre for Physical Activity Research (CFAS), Copenhagen
  - Rigshospitalet, Copenhagen

IPD SHARING:
Plan to Share IPD: Yes
The data will be openly available in a repository.
Supporting Information: Study Protocol, SAP, Analytic Code